CLINICAL TRIAL: NCT01274520
Title: Hypothermic Machine Preservation of Extended Criteria Liver Allografts for Transplantation
Brief Title: Hypothermic Machine Preservation-Phase 2
Acronym: HMP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD6236
Record Dates: First submitted 2010-11-03; First posted 2011-01-11 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Liver Damage
Keywords: ECD liver transplant allografts; Hypothermic machine perfusion; Cold storage preservation; liver transplant; portable bypass system; machine perfusion preservation; extended criteria liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental: Hypothermic Machine Perfusion Group (Experimental): The Medtronic Portable Bypass System (PBS®) with Model 550 Bioconsole and the BioCal® blood temperature control module will be used for machine perfusion of liver grafts. These products are commercially available and used in clinical practice for cardiopulmonary bypass and extracorporeal membrane oxygenation. The Medtronic system utilizes an atraumatic centrifugal pump that can deliver the flow rates approximating portal venous flow in human livers, and it has modules for online membrane oxygenation, and electronic flow measurement.
  Interventions: Device: The Medtronic Portable Bypass System (PBS®)
- Matched control group (No Intervention): The proposed study is a matched cohort design. Subjects will be matched with 24 historical control patients who received similar cold stored ECD grafts. Subjects will be matched on known covariates including donor age, donation after cardiac death, steatosis, both warm and cold ischemia times, recipient age, MELD score and disease etiology. Additional analyses will be performed on historical control blood and/or tissue samples previously collected and stored in the study's sample repository.

INTERVENTIONS:
Device: The Medtronic Portable Bypass System (PBS®) — Will be used for machine perfusion of liver grafts.
  Other Names: Medtronic Portable Bypass System (PBS®)
  Arms: Experimental: Hypothermic Machine Perfusion Group

SUMMARY:
This is a study comparing a technique of continuous circulation to the liver as a means of preventing liver damage during transportation to the transplant hospital. This new technique of Machine Perfusion (MP) will be compared to the standard technique where the liver is maintained in a bag of solution on ice without circulation. The investigators will evaluate and compare the outcomes of the transplants with the new technique to the standard technique. There will be 24 MP patient's in the study. The investigators have previously used this technique with success in 20 human liver transplant patients. The investigators think there will be a benefit in terms of less damage to and better function of the donor liver which will result in faster recovery for the patients. This protective effect may allow us to successfully transplant more patients and prevent people from dying while waiting for a liver transplant.

DETAILED DESCRIPTION:
It is our hypothesis that liver machine perfusion will increase the safe utilization of the existing supply of extended criteria donor (ECD) livers by (1) increasing the quality and duration of preservation thereby reducing the clinical effects reperfusion injury (2) improving early outcomes in patients receiving ECD liver allografts (3) developing reliable markers for pretransplant assessment of the potential graft (4) giving surgeons more confidence when transplanting ECD livers and (5) allowing an avenue for ex vivo manipulation of the liver to protect or restore a transiently injured liver.

The proposed study is a matched cohort design. Potential subjects will be recruited from the Center for Liver Disease and Transplantation (CLDT) active Liver Transplant Waiting List. The Principal Investigator as well as the CoInvestigators, are all actively involved in the pre transplant evaluation process. Patients who are on the Waiting List and have provided written consent to receive an ECD graft will be recruited for this trial. Subjects will be matched with 24 historical control patients who received similar cold stored ECD grafts. Subjects will be matched on known covariates including donor age, donation after cardiac death, steatosis, both warm and cold ischemia times, recipient age, Model End-Stage Liver Disease (MELD) score and disease etiology.

Subjects will be noncritically ill, not in an intensive care unit, and have a MELD < 35 in order to minimize the variability in outcome in the sickest patients. All subjects must provide written informed consent and meet the inclusion and exclusion criteria.

Subjects will be followed for one year post transplantation, in conjunction with their routine liver transplant followup appointments. Retention of subjects for this trial will not be a challenge, in that the followup visit time points (postoperative days 1 through the discharge date, 7, 14, 30, 90, 180 and 365) are all consistent with our standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed IRB consent by patient or patient's legally appointed representative.
* Be at least 18 years of age; male or female.
* Listed with UNOS for liver transplantation.
* Organ declined by at least one transplant center
* Extended criteria donor as defined by:

  * Presence of hepatitis C antibody
  * Donation after Cardiac Death (DCD)
  * Severe Hypernatremia: donor serum sodium >165 meq/L for at least 12 hours prior to procurement
  * Donor age ≥65 years
  * Presence of significant steatosis >25% macrovesicular by biopsy
  * Evidence of significant donor ischemic injury
  * Current donor serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1000 IU/L
  * Ischemic injury evidenced by prolonged hypotension, high pressor requirement and/or rising serum liver function tests or one test more than five times the upper limit of normal (AST, ALT, or Total Bilirubin)

Exclusion Criteria:

* Patients in whom the donor liver will be subjected to less than 4 hours of cold ischemia (surgeon desires immediate implantation)
* Patient hospitalized in intensive care unit (ICU) at time of transplantation and/or physiologic MELD score >35
* Dual organ recipient
* ABO incompatibility
* Retransplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12-19 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V Guarrera, MD, FACS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guarrera JV, Henry SD, Samstein B, Reznik E, Musat C, Lukose TI, Ratner LE, Brown RS Jr, Kato T, Emond JC. Hypothermic machine preservation facilitates successful transplantation of "orphan" extended criteria donor livers. Am J Transplant. 2015 Jan;15(1):161-9. doi: 10.1111/ajt.12958. Epub 2014 Dec 17. PMID 25521639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 liver recipients who received extended criteria donor (ECD) liver transplant allografts were recruited for our treatment group over a span of 2 years. As a high-volume, major NY transplant center with approximately 270 adult patients on our Liver Transplant Waiting List and 45-50% receiving ECD grafts, we were able to meet our enrollment goal.
Groups:
- Matched Control Group: This study had a matched cohort design. Treatment subjects were matched with 25 historical control patients who received similar cold stored ECD grafts. Subjects were matched on known covariates including donor age, donation after cardiac death, steatosis, both warm and cold ischemia times, recipient age, MELD score and disease etiology. Additional analyses were performed on historical control blood and/or tissue samples previously collected and stored in the study's sample repository.
- Experimental: Medtronic Portable Bypass System Group: 24 subjects were treated with the Medtronic Portable Bypass System (PBS®) with Model 550 Bioconsole, and the BioCal® blood temperature control module was used for machine perfusion of liver grafts. These products are commercially available and are used in clinical practice for cardiopulmonary bypass and extracorporeal membrane oxygenation. The Medtronic system utilizes an atraumatic centrifugal pump that can deliver the flow rates approximating portal venous flow in human livers, and it has modules for online membrane oxygenation, and electronic flow measurement.
Period: Overall Study
Arm/Group | Matched Control Group | Experimental: Medtronic Portable Bypass System Group
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Experimental group: Adult recipients of ECD deceased donor liver grafts (organ must have been declined by ≥1 transplant center) who were non-critically ill (not in intensive care, MELD < 35) at time of transplant.
  Historical control group: Patients who received liver grafts with similar donor characteristics and standard cold storage preservation.
Groups:
- Matched Control Group: This study had a matched cohort design. Treatment subjects were matched with 25 historical control patients who received similar cold stored extended criteria donor (ECD) grafts. Subjects were matched on known covariates including donor age, donation after cardiac death, steatosis, both warm and cold ischemia times, recipient age, Model for End-Stage Liver Disease (MELD) score and disease etiology. Additional analyses were performed on historical control blood and/or tissue samples previously collected and stored in the study's sample repository.
- Experimental: Hypothermic Machine Perfusion Group Group: 24 subjects were treated with the Medtronic Portable Bypass System (PBS®) with Model 550 Bioconsole, and the BioCal® blood temperature control module was used for machine perfusion of liver grafts. These products are commercially available and are used in clinical practice for cardiopulmonary bypass and extracorporeal membrane oxygenation. The Medtronic system utilizes an atraumatic centrifugal pump that can deliver the flow rates approximating portal venous flow in human livers, and it has modules for online membrane oxygenation, and electronic flow measurement.
- Total: Total of all reporting groups
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group Group | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Customized [Number; unit: participants]
  18-21 years | 0 | 0 | 0
  22-29 years | 0 | 0 | 0
  30-39 years | 0 | 1 | 1
  40-49 years | 3 | 3 | 6
  50-59 years | 11 | 9 | 20
  60-69 years | 8 | 9 | 17
  70-79 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 3 | 14
  Not Hispanic or Latino | 13 | 18 | 31
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Number; unit: participants] — Racial Category (Single category per participant)
  participants
    White | 16 | 14 | 30
    Black or African American | 7 | 5 | 12
    Multiracial | 0 | 0 | 0
    Other | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival at One Year Post-Transplantation
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: participants
Groups:
- Matched Control Group: This study had a matched cohort design. Treatment subjects were matched with 25 historical control patients who received similar cold stored extended donor criteria (ECD) grafts. Subjects were matched on known covariates including donor age, donation after cardiac death, steatosis, both warm and cold ischemia times, recipient age, MELD score and disease etiology. Additional analyses were performed on historical control blood and/or tissue samples previously collected and stored in the study's sample repository.
- Experimental: Hypothermic Machine Perfusion Group: 24 subjects were treated with the Medtronic Portable Bypass System (PBS®) with Model 550 Bioconsole, and the BioCal® blood temperature control module was used for machine perfusion of liver grafts. These products are commercially available and are used in clinical practice for cardiopulmonary bypass and extracorporeal membrane oxygenation. The Medtronic system utilizes an atraumatic centrifugal pump that can deliver the flow rates approximating portal venous flow in human livers, and it has modules for online membrane oxygenation, and electronic flow measurement.
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
participants | 19 | 19

2. Primary Outcome: Graft Survival at One Year Post-Transplantation
Description: Analysis was based on the amount of liver allografts in each cohort that were deemed to be clinically functional at 1 year post-transplantation (i.e. no re-transplantation required).
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: grafts
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
grafts | 23 | 23

3. Secondary Outcome: Incidence of Primary Graft Nonfunction
Description: Incidence of Primary Graft Nonfunction (PNF), defined as follows:
  * Relisted for orthotopic liver transplantation (OLT) within 7 days of OLT, not for vascular thromboses
  * Alanine aminotransferase (ALT) >2000 and one or both of: acidosis with pH <7.3 or lactate >2X (two times) normal
  * International normalized ratio (INR) >2.5
Time Frame: Post-Operative Day 1 to Day 7
Measure: Number; unit: participants
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
participants | 2 | 1

4. Secondary Outcome: Incidence of Early Allograft Dysfunction (EAD)
Description: Incidence of Early Allograft Dysfunction (EAD), defined as follows:
  * Bilirubin >10 on post-operative day (POD)#7
  * International normalized ratio (INR) >1.6 on POD#7
  * Transaminase level (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) >2000 within the first 7 days
Time Frame: Within the first 7 days post-transplantation
Measure: Number; unit: participants
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
participants | 9 | 5

5. Secondary Outcome: Incidence of Post-Operative Complications
Description: Incidence of Retransplants or Hepatic Artery Thrombosis (HAT) within 1 month post-transplantation
Time Frame: 1 Month Post-Transplantation
Measure: Number; unit: participants
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
participants
  Retransplant | 0 | 1
  HAT | 1 | 1

6. Secondary Outcome: Incidence of Bile Leaks
Description: Incidence of bile leaks.
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: events
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
events | 3 | 0

7. Secondary Outcome: Incidence of Re-Operation For Bleeding
Description: Incidence of patients who required re-operation for a bleeding event
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: participants
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
participants | 5 | 2

8. Secondary Outcome: Incidence of Hernia Events Within 1 Year Post-Transplantation
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: hernia events
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
hernia events | 2 | 4

9. Secondary Outcome: Hospital Length of Stay (Index Transplant Hospitalization)
Description: Length of transplant hospital stay post-transplantation (Index Transplant Hospitalization)
Time Frame: First admission after transplant
Measure: Mean (Full Range); unit: days
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
days | 16.5 [7 to 52] | 10 [6 to 51]

10. Secondary Outcome: Time With Stent (Days)
Description: Measure of biliary complications as evidenced by mean time with stent (in days).
Time Frame: Post-Operative Day 1 to Day 365
Measure: Mean (Full Range); unit: days
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group Group
Number analyzed (Participants) | 25 | 24
days | 86 [14 to 365] | 66.5 [54 to 79]

11. Secondary Outcome: Incidence of Biliary Strictures
Description: Incidence of biliary strictures.
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: events
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
events | 10 | 2

12. Secondary Outcome: Incidence of Endoscopic Retrograde Cholangiopancreatographies (ERCPs)
Description: Incidence of endoscopic retrograde cholangiopancreatographies (ERCPs)
Time Frame: Post-Operative Day 1 to Day 365
Measure: Number; unit: events
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group
Number analyzed (Participants) | 25 | 24
events | 35 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious Adverse Event (SAE) is defined as any clinically significant event which required a hospitalization admission during the subject's participation in the trial. Only SAEs were reported for the purposes of data collection and data analysis in this study.
Arm/Group | Matched Control Group | Experimental: Hypothermic Machine Perfusion Group Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 6/24
Serious Adverse Events (participants affected / at risk) | 11/25 | 6/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Control Group (N=25) | Experimental: Hypothermic Machine Perfusion Group Group (N=24)
Events Requiring Hospitalization (Hepatobiliary disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes